CLINICAL TRIAL: NCT04497194
Title: Registry of Biological Samples, Clinical Information and Epidemiological Data of COVID-19 Patients Admitted at the University Hospital of Verona (AOUI Verona)
Brief Title: Registry of COVID-19 Patients at AOUI Verona
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Evelina Tacconelli, Professor, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: COVID19-VR
Record Dates: First submitted 2020-05-18; First posted 2020-08-04 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: not applicable (observational study) — not applicable (observational study)

SUMMARY:
The registry of COVID-19 patients was designed to collect epidemiolgical, demographic, clinical, anamnestic and outcome information together with serological and microbiological samples from COVID-19 patients admitted at the University Hospital of Verona (Azienda Ospedaliera Universitaria Integrata, AOUI Verona). All SARS-CoV 2 positive patients admitted and able to give an informed consent are included, irrespectively of age and gender.

DETAILED DESCRIPTION:
Anamnestic data are collected at the enrollment, while all the other clinical and epidemiological information are retrieved retrospectively from patients' medical records and electronic health records.

Serological and microbiological samples (blood samples, fecal samples and nasal/rectal swabs) are collected within 48 hours after admission and during the hospital stay, according with routine internal procedures.The biological samples are stored at the University Laboratory for Medical Research (Laboratorio Universitario di Ricerca Medica, LURM).

A dedicated database has been created and implemented to collect all the above mentioned information.

ELIGIBILITY:
Inclusion Criteria:

* PCR for SARS-CoV 2 positive on NPS swab or high suspicion of SARS-CoV 2 with ongoing swab;
* All ages;
* All genders;
* Informed consent obtained.

Exclusion Criteria:

* Failure to obtain the informed consent.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: COVID-19 patients admitted at the University Hospital of Verona (Azienda Ospedaliera Universitaria Integrata, AOUI Verona).
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Epidemiological predictors of poor outcomes in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  Epidemiological data including demographic data, contact with COVD-19 positive patients and onset of symptoms.
Clinical predictors of poor outcomes in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  Underlying chronic diseases, signs/symptoms related with COVID-19 diseases an clinical presentation on admission
Body temperature (°C) on admission in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  Body temperature (°C)
Blood pressure (mmHg) on admission in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  Blood pressure (mmHg)
Pulse rate (beats per minute) on admission in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  Pulse rate (beats per minute)
Respiratory rate (breaths per minute) on admission in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  Pulse rate (beats per minute)
Peripheral oxygen saturation (%) on admission in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  Peripheral oxygen saturation (%)
C reactive protein (CRP, m/gL) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  CRP (m/gL)
Procalcitonin (PCT, ng/mL) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  PCT (ng/mL
White Blood Count (WBC, cell/mm3) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  White Blood Count (WBC, cell/mm3)
Neutrophils (cell/mm3) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  Neutrophils (cell/mm3)
Lymphocytes (cell/mm3) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  Lymphocytes (cell/mm3)
Platelets (cell/mm3) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  Platelets (cell/mm3)
L-lattato deidrogenasi (LDH, mU/ml) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  LDH (mU/ml)
Creatine kinase (CK, U/L) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  CK (U/L)
D-dimer (μg/L) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  D-dimer (μg/L)
fibrinogen (g/L) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  fibrinogen (g/L)
ferritin (mcg/L) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  ferritin (mcg/L)
AST (U/L) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  AST (U/L)
ALT (U/L) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  ALT (U/L)
Creatinine (mg/dl) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  Creatinine (mg/dl)
Arterial blood gas anaysis pH in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  pH
Arterial blood gas anaysis pO2 (mmHg) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  pO2 (mmHg)
Arterial blood gas anaysis pCO2 (mmHg) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  pCO2 (mmHg)
Arterial blood gas anaysis HCO3 (mmol/l) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  HCO3 (mmol/l)
Arterial blood gas anaysis SpO2 (%) in COVID-19 patients admitted to University Hospital of Verona | through study completion, an average of 3 months
  SpO2 (%)
Host-related factors associated with the pathogenesis of COVID-19 | through study completion, an average of 3 months
  IL-6 (pg/mL)
Virological factors associated with the pathogenesis of COVID-19 | through study completion, an average of 3 months
  Nasal and rectal swabs, fecal samples and blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided